CLINICAL TRIAL: NCT01120236
Title: A Randomized Phase II Study of Androgen Deprivation Combined With IMC-A12 Versus Androgen Deprivation Alone for Patients With New Hormone Sensitive Metastatic Prostate Cancer
Brief Title: Bicalutamide and Goserelin or Leuprolide Acetate With or Without Cixutumumab in Treating Patients With Newly Diagnosed Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02003; NCI-2011-02003 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0925; CDR0000663832; S0925 (Other: SWOG); S0925 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; cixutumumab; Goserelin; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (androgen deprivation and cixutumumab) (Experimental): Patients receive androgen deprivation therapy comprising bicalutamide PO QD on days 1-28 and either goserelin acetate SC or leuprolide acetate IM every 1, 3, 4, 6, or 12 months. Patients also receive cixutumumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Biological: Cixutumumab; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Other: Pharmacological Study
- Arm II (androgen deprivation therapy) (Active Comparator): Patients receive androgen deprivation therapy comprising bicalutamide and either goserelin acetate or leuprolide acetate as in arm I.
  Interventions: Drug: Bicalutamide; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Other: Pharmacological Study

INTERVENTIONS:
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
  Arms: Arm I (androgen deprivation and cixutumumab)
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial is studying bicalutamide, goserelin, or leuprolide acetate to see how well they work when given with or without cixutumumab in treating patients with newly diagnosed metastatic prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, goserelin, or leuprolide acetate, may lessen the amount of androgens made by the body. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether bicalutamide, goserelin, or leuprolide acetate are more effective when given with or without cixutumumab in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the undetectable prostate-specific antigen (PSA) rate (PSA < 0.2 ng/mL) after seven cycles (28 weeks) of protocol treatment between those randomized to a luteinizing hormone-releasing hormone (LHRH) agonist and bicalutamide and those randomized to a LHRH agonist, bicalutamide and IMC-A12 (cixutumumab).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of IMC-A12 with a LHRH agonist and bicalutamide.

II. To compare the proportion of men who do not achieve a PSA of < 4 ng/mL between the two groups.

III. To assess the accuracy of the prognostic model of undetectable PSA that was developed from Southwest Oncology Group (SWOG)-9346 using current trial data from each arm.

IV. To assess serum samples and peripheral blood mononuclear cells (PBMNC) for pharmacodynamic activity with potential biomarkers for IMC-A12 (including, but not limited to: insulin-like growth factor [IGF]-I, free IGF-I, IGF-II, IGF binding protein [IGFBP]2, IGFBP3, growth hormone, insulin and C-peptide) obtained from optional blood specimens both before initiation of androgen deprivation therapy and twelve weeks after initiation of combined therapy.

V. To determine baseline pre-treatment circulating tumor cell (CTC) quantities and response to therapy (for those patients with detectable CTC levels >= 1) twelve weeks later.

VI. In the same subset of patients where CTC levels are obtained, determine baseline serum levels of micro-ribonucleic acids (RNAs) to include but not limited to microRNA (mi)-141 both before initiation of androgen deprivation therapy and twelve weeks after combined therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive androgen deprivation therapy comprising bicalutamide orally (PO) once daily (QD) on days 1-28 and either goserelin acetate subcutaneously (SC) or leuprolide acetate intramuscularly (IM) every 1, 3, 4, 6, or 12 months. Patients also receive cixutumumab intravenously (IV) over 1 hour on days 1 and 15. Treatment repeats every 28 days for 7 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive androgen deprivation therapy comprising bicalutamide and either goserelin acetate or leuprolide acetate as in arm I.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologically or cytologically proven diagnosis of adenocarcinoma of the prostate; note: If there is no formal biopsy report documenting the diagnosis of prostate cancer, the patient can be allowed on trial if the PSA level is at least 20, and there are at least three definitive metastatic lesions seen on scan; all patients must have had metastatic (M1) disease as evidenced by soft tissue and/or bony metastases prior to androgen deprivation therapy initiation; patients must have at least one of the following at the time they started androgen deprivation therapy:

  * Visceral disease (liver, lung, or other viscera)
  * Bone metastases to sites in either the axial (spine, pelvis, ribs, or skull) and/or the appendicular (clavicle, humerus, or femur) skeleton
  * Lymph node disease not considered to be encompassed within a single radiotherapy port (e.g., above the aortic bifurcation, etc.)
* Patients who have measurable disease must have radiographic assessment (at least an abdominal/pelvic computed tomography [CT]) within 28 days prior to registration; non-measurable disease must also be assessed (e.g., bone scan) in all patients within 56 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients must have a PSA >= 5 ng/mL obtained within 90 days prior to initiation of androgen deprivation therapy
* Patients with known brain metastases are not eligible; brain imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms, but if brain imaging studies are performed, they must be negative for disease
* Patient must have had no more than 30 days of prior medical castration for metastatic prostate cancer (prior androgen deprivation therapy is allowed if it was received with curative intent in the neoadjuvant, concurrent, and/or adjuvant fashion and at least 2 years have elapsed since completion of androgen deprivation therapy); the start date of medical castration is considered the day the patient first received an injection of a LHRH agonist, not an oral antiandrogen; if the method of castration is luteinizing hormone releasing hormone (LHRH) agonists (i.e., leuprolide or goserelin), the patient must be willing to continue the use of LHRH agonists and add bicalutamide for combined androgen deprivation therapy (ADT) during protocol treatment; the 30 day window begins from the date of receiving the LHRH agonist, not the oral antiandrogen; if the patient was on a different antiandrogen (e.g. flutamide), the patient must be willing to switch over to bicalutamide; patients must not have received bilateral orchiectomy; patients must not have received or be planning to receive LHRH antagonists (i.e., Degarelix); however, if the patient was initiated on a LHRH antagonist within the 30 day window and is willing to switch to a LHRH agonist with bicalutamide, he may enroll on the late induction group
* Patients who have not already started androgen deprivation therapy must be offered the opportunity to participate in the translational medicine studies; once a patient has started any form of antiandrogen (i.e., either bicalutamide or LHRH agonist), he is not eligible for any translational medicine studies
* Patients must not have received any prior cytotoxic chemotherapy for metastatic prostate cancer; prior cytotoxic chemotherapy with curative intent in the neoadjuvant or adjuvant setting is allowed; patients must not have received any prior treatment with agents that directly inhibit IGF or IGFRs
* Patients must not have received prior strontium-89, rhenium-186, rhenium-188, or samarium-153 radionuclide therapy within 28 days prior to registration
* Patients may have received prior radiation therapy or biologic therapy (e.g. vaccines, immunotherapy, anti-sense, small molecules, monoclonal antibodies); however, at least 28 days must have elapsed since completion of therapy and patient must have recovered from all side effects
* Patients may have received prior surgery; for all major surgeries, at least 28 days must have elapsed since completion and patient must have recovered from all side effects
* Leukocytes >= 3,000 mcL
* Absolute neutrophil count (ANC) >= 1,500 mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Bilirubin =< 1.5 times the institutional upper limit of normal (ULN) (unless documented Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 times the institutional ULN, or =< 5 times the institutional ULN if liver metastases are present
* Creatinine =< 2.0 x the institutional ULN or calculated creatinine clearance >= 40 mL/min
* International normalized ratio (INR) =< 1.5
* Partial thromboplastin time (PTT) no more than 5 seconds above the institutional ULN
* Patients receiving prophylactic low dose coumadin or low molecular weight heparin are eligible as long as they meet these coagulation criteria; patients requiring full-dose (therapeutic) anticoagulation are eligible provided that they have been on a stable dose of anticoagulation and the coagulation parameters are stable within the therapeutic range (e.g., INR 2-3 for patients on therapeutic warfarin)
* Patients must have a hemoglobin A1c (HgA1c) =< 7% AND fasting glucose of < 160 mg/dL or below the institutional ULN within 14 days prior to registration; patients with diabetes mellitus who meet this criterion must be on a stable dietary or therapeutic regimen for this condition
* Patients must not have a history of symptomatic congestive heart failure or a known ejection fraction (left ventricular ejection fraction [LVEF]) that is >= 10% below the lower limit of normal (LLN); if left ventricular (LV) dysfunction is suspected, but not confirmed by review of past medical history, a multi gated acquisition scan (MUGA) or echocardiogram must be obtained within 90 days prior to registration
* Patient must not have a history of allergic reaction attributed to compounds of similar chemical or biologic composition to IMC-A12; patients must not have received prior chimerized or murine monoclonal antibody therapy
* Patients must have a Zubrod performance status of 0 - 2; Zubrod performance status 3 will be allowed if from bone pain only
* Patients with human immunodeficiency virus (HIV) positivity requiring antiretroviral therapy are not eligible for this study
* Patients must have no plans to receive concurrent chemotherapy, hormonal therapy (other than the LHRH agonist and oral anti-androgen), radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol treatment; concurrent bone targeting agents that do not have effect on PSA (i.e. denosumab or zoledronic acid) are allowed
* Patients must have no plans to receive concurrent five-alpha reductase inhibitors (e.g. finasteride and dutasteride), ketoconazole, diethylstilbestrol/DES, or other estrogen-based therapy while on this protocol treatment
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Men of reproductive potential must have agreed to use an effective contraceptive method while receiving treatment on this study and for at least three months after protocol treatment ends
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As part of the OPEN registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Yu, Principal Investigator — SWOG Cancer Research Network
Locations (170):
- United States (169):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Tahoe Forest Cancer Center, Truckee, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Reid Health, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - University of Rochester, Rochester, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Saint Charles Medical Center-Bend, Bend, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Yu EY, Li H, Higano CS, Agarwal N, Pal SK, Alva A, Heath EI, Lam ET, Gupta S, Lilly MB, Inoue Y, Chi KN, Vogelzang NJ, Quinn DI, Cheng HH, Plymate SR, Hussain M, Tangen CM, Thompson IM Jr. SWOG S0925: A Randomized Phase II Study of Androgen Deprivation Combined With Cixutumumab Versus Androgen Deprivation Alone in Patients With New Metastatic Hormone-Sensitive Prostate Cancer. J Clin Oncol. 2015 May 10;33(14):1601-8. doi: 10.1200/JCO.2014.59.4127. Epub 2015 Apr 6. PMID 25847934

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Started | 105 | 106
Ineligble | 0 | 1 (Patient ineligible due to no demonstable radiographic metastasis and is excluded from all analyses.)
Completed | 105 | 105
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient from Arm II (androgen deprivation therapy) was ineligible because of lack of a demonstrable radiographic metastasis. This patient was excluded from analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy) | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [60 to 72] | 66 [58 to 73] | 66 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 105 | 105 | 210
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 4 | 10 | 14
  White | 94 | 88 | 182
  Other | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 105 | 105 | 210
Prostate-Specific Antigen (PSA) [Median (Inter-Quartile Range); unit: ng/mL] | 31 [12 to 74] | 37 [10 to 200] | 34 [11 to 133]
Weight [Median (Inter-Quartile Range); unit: kg] | 90 [79 to 101] | 86 [77 to 98] | 88 [77 to 100]
Body Mass Index (BMI) [Number; unit: participants]
  <18.5 (underweight) | 1 | 2 | 3
  18.5 to 24.9 (normal weight) | 21 | 29 | 50
  25 to 29.9 (overweight) | 36 | 39 | 75
  >= 30 (obese) | 43 | 33 | 76
  Unknown | 4 | 2 | 6
Gleason Score [Number; unit: participants] — This is a 2 to 10 grading system for prostate carcinoma devised by Dr. Donald Gleason in 1977 as a method for predicting the behavior of prostate cancer. Tumors with a low Gleason score are less likely to show aggressive behavior and therefore are less likely to have spread outside of the gland to lymph nodes. To obtain a Gleason score, the dominant tumor pattern is added to the second most prevalent pattern to obtain a number between 2 and 10. If a tumor has patterns 3 and 2, the score would be 5. If the tumor has only one pattern, then the single pattern is added to itself (e.g. 3+3=6).
  participants
    <7 | 8 | 6 | 14
    7 | 29 | 11 | 40
    >=7 | 63 | 82 | 145
    Unknown | 5 | 6 | 11
Zubrod Performance Score [Number; unit: participants] — Scale 0 (best) to 2 (worst)
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. = Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  participants
    0 | 62 | 65 | 127
    1 | 41 | 38 | 79
    2 | 2 | 2 | 4
Site of Metastasis [Number; unit: participants]
  Lymph Node Only | 15 | 9 | 24
  Bone Only | 56 | 63 | 119
  Lymph Node and Bone | 19 | 17 | 36
  Visceral | 15 | 16 | 31
Bone Pain [Number; unit: participants] | 28 | 35 | 63
Early Induction Androgen Deprivation [Number; unit: participants] — Prior remote AD was allowed only if received in the neoadjuvant, concurrent, and/or adjuvant settings and > 2 years had elapsed since completion of therapy.
  participants | 59 | 65 | 124

OUTCOME MEASURES:

1. Primary Outcome: Undetectable PSA Rate
Description: Undetectable PSA rate (<= 0.2 ng/mL) after seven cycles (28 weeks) of protocol treatment
Time Frame: 7 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 105 | 105
participants | 42 | 34
Statistical Analysis 1: Comparison: Arm I (Androgen Deprivation and Cixutumumab) vs Arm II (Androgen Deprivation Therapy); An intention-to-treat approach was used in analysis of the primary endpoint. A 45% undetectable PSA <= 0.2 ng/mL rate at 28 weeks was assumed for (control) arm II , based on data from SWOG 9346. Using a one-sided type I error rate of 0.10, we had 90% statistical power to detect an absolute difference of 20% in the undetectable PSA rate with the addition of cixutumumab using Fisher's exact test; Test type: Superiority or Other; p = 0.16, Fisher Exact; Risk Ratio (RR) = 1.24 — Arm I (Androgen Deprivation and Cixutumumab) represents the numerator and Arm II (Androgen Deprivation Therapy) represents the denominator for relative risk

2. Secondary Outcome: Toxicity
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 28 weeks
Population: All participants receiving at least some protocol treatment were included in toxicity analysis. Four patients on Arm I (androgen deprivation and cixutumumab) and two patients on Arm II (androgen deprivation therapy) did not receive any protocol treatment and were therefore excluded from this analysis.
Measure: Number; unit: Participants
Groups:
- Arm I (Androgen Deprivation and Cixutumumab): Patients receive androgen deprivation therapy comprising bicalutamide PO QD on days 1-28 and either goserelin acetate SC or leuprolide acetate IM every 1, 3, 4, 6, or 12 months. Patients also receive cixutumumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for 7 courses in the absence of disease progression or unacceptable toxicity.
  Bicalutamide: Given PO Cixutumumab: Given IV Goserelin Acetate: Given SC Laboratory Biomarker Analysis: Correlative studies Leuprolide Acetate: Given IM Pharmacological Study: Correlative studies
- Arm II (Androgen Deprivation Therapy): Patients receive androgen deprivation therapy comprising bicalutamide and either goserelin acetate or leuprolide acetate as in arm I.
  Bicalutamide: Given PO Goserelin Acetate: Given SC Laboratory Biomarker Analysis: Correlative studies Leuprolide Acetate: Given IM Pharmacological Study: Correlative studies
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 101 | 104
Participants
  Alanine aminotransferase increased | 1 | 0
  Anemia | 1 | 1
  Anxiety | 0 | 1
  Aspartate aminotransferase increased | 1 | 0
  Cognitive disturbance | 1 | 0
  Depression | 0 | 1
  Erectile dysfunction | 1 | 0
  Exostosis | 1 | 0
  Glucose intolerance | 0 | 1
  Hot flashes | 1 | 1
  Hypercalcemia | 2 | 0
  Hyperglycemia | 8 | 0
  Hypertension | 2 | 2
  Hypertriglyceridemia | 1 | 0
  Left ventricular systolic dysfunction | 1 | 0
  Nausea | 1 | 0
  Obesity | 1 | 1
  Soft tissue infection | 1 | 0
  Urinary tract infection | 1 | 0
  Urinary tract obstruction | 0 | 1
  Vomiting | 1 | 0

3. Secondary Outcome: Proportion of Patients Who do Not Achieve a Partial PSA Response
Description: A partial PSA response is considered <= 4 ng/mL
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 105 | 105
participants | 46 | 56
Statistical Analysis 1: Comparison: Arm I (Androgen Deprivation and Cixutumumab) vs Arm II (Androgen Deprivation Therapy); Proportion of patients in each arm with PSA > 4 ng/mL after seven cycles of protocol treatment were compared; Test type: Superiority or Other; p = 0.11, Fisher Exact; Risk Ratio (RR) = 0.82 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Accuracy of the Prognostic Model of Undetectable PSA (Developed From SWOG-9346)
Description: The logistic regression algorithm for predicting undetectable PSA that was developed for SWOG-9346 using its baseline risk factors (age at registration, performance status, baseline PSA, and bone pain) will be applied to each arm of this trial to evaluate the level of agreement between the observed and predicted undetectable PSA rates.
Time Frame: Up to 5 years
Population: The data from this trial was intended to be used as a validation dataset for the prognostic model built using data from SWOG-9346. However, data for this objective was not collected.
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Correlation of microRNA Measures With 28-week PSA Response
Description: The Friedman test will be used to evaluate correlations between microRNA measures (CT) and 28-week PSA response.
Time Frame: Baseline to 28 weeks
Population: Among the 50 patients in this biomarker substudy, 10 patients were excluded: 1 ineligible for S0925, 6 started LHRH therapy prior to registration, 3 had insufficient miRNA samples. The remaining 40 patienets were included in this analysis.
Measure: Median (Full Range); unit: Cycle Threshold (CT)
Groups:
- PSA Complete Response: Patients who had a PSA level of ≤ 0.2 ng/mL at 28 weeks after registration, pooled treatment Arm I (androgen deprivation and cixutumumab) & Arm II (androgen deprivation therapy)
- PSA Partial Response: Patients who had a PSA level of >0.2 ng/mL and <= 4.0 ng/mL at 28 weeks after registration, pooled treatment Arm I (androgen deprivation and cixutumumab) & Arm II (androgen deprivation therapy)
- PSA Non-Responders: Patients who had a PSA level of > 4.0 ng/mL at 28 weeks after registration, pooled treatment Arm I (androgen deprivation and cixutumumab) & Arm II (androgen deprivation therapy)
Arm/Group | PSA Complete Response | PSA Partial Response | PSA Non-Responders
Number analyzed (Participants) | 22 | 5 | 13
Cycle Threshold (CT)
  miR-141 | 32.6 [29.5 to 36.8] | 32.0 [31.9 to 32.7] | 31.5 [27.6 to 33.5]
  miR-200a | 34.5 [31.4 to 39.9] | 33.8 [32.4 to 35.6] | 33.8 [30.1 to 40.0]
  miR-200b | 33.6 [32.7 to 35.0] | 33.6 [32.7 to 35.0] | 32.6 [29.3 to 34.8]
  miR-210 | 32.5 [30.8 to 36.8] | 32.1 [31.3 to 33.8] | 32.3 [28.0 to 34.3]
  miR-375 | 33.0 [29.3 to 35.9] | 32.6 [30.0 to 35.0] | 29.5 [25.7 to 33.8]

6. Secondary Outcome: Correlation of microRNA Measures With Baseline Circulating Tumor Cell (CTC) Counts
Description: The Friedman test will be used to evaluate correlations between microRNA measures (CT) and Baseline CTCs.
Time Frame: Baseline
Population: Among the 50 patients in this biomarker substudy, 14 patients were excluded: 1 ineligible for S0925, 6 started LHRH therapy prior to registration, 3 had insufficient miRNA samples and 4 had insufficient CTC samples. The remaining 36 patients were used in this analysis.
Measure: Median (Full Range); unit: Cycle Threshold (CT)
Groups:
- CTC=0: No CTCs foundin 7.5 mL blood sample collected at baseline, pooled treatment arms
- CTC= 1-4: 1 to 4 CTCs found in 7.5 mL blood sample collected at baseline, pooled treatment arms
- CTC= 5+: Five or more CTCs were found in 7.5 mL blood sample collected at baseline, pooled treatment arms
Arm/Group | CTC=0 | CTC= 1-4 | CTC= 5+
Number analyzed (Participants) | 14 | 8 | 14
Cycle Threshold (CT)
  miR-141 | 33.0 [31.5 to 36.8] | 32.7 [31.6 to 33.7] | 31.9 [28.8 to 32.5]
  miR-200a | 34.4 [31.4 to 39.7] | 34.7 [32.1 to 37.7] | 33.0 [30.1 to 40.0]
  miR-200b | 33.4 [32.1 to 34.2] | 33.2 [32.7 to 34.1] | 33.6 [29.3 to 35.0]
  miR-210 | 32.5 [30.8 to 36.8] | 32.7 [31.4 to 34.3] | 32.1 [31.0 to 33.5]
  miR-375 | 32.8 [30.1 to 35.1] | 32.7 [26.5 to 35.9] | 30.2 [26.7 to 35.0]

7. Secondary Outcome: Change in Level of CTCs
Description: Will be correlated with 28-week PSA response.
Time Frame: Baseline to 28 weeks
Population: Among the 50 patients in this biomarker substudy, 1 was ineligible for the trial, 6 started LHRH therapy prior to registration, and 4 had CTC blood samples that were not assay evaluable. The remaining 39 patients were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CTC=0 | CTC= 1-4 | CTC= 5+
Number analyzed (Participants) | 16 | 9 | 14
Participants
  PSA <= 0.2 ng/mL | 12 | 5 | 4
  0.2 < PSA <=4.0 ng/mL | 0 | 2 | 3
  PSA > 4.0 ng/mL | 4 | 2 | 7

8. Other Pre Specified Outcome: Change in Level of IGF-I, Free IGF-I and C-peptide
Description: Serum samples and peripheral blood mononuclear cells (PBMNC) for pharmacodynamic activity with potential biomarkers for IMC-A12 (including, but not limited to: IGF-I, free IGF-I and C-peptide) obtained from optional blood specimens both before initiation of androgen deprivation therapy and twelve weeks after initiation of combined therapy. Results are reported as the difference between baseline and 12 weeks after start of therapy.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 18 | 9
ng/mL
  C-peptide | -7 (24.5) | 3 (20.1)
  IGF-I | 0 (2.4) | 1 (2.7)
  IGF-II | 10 (46.7) | -6 (43.7)

9. Other Pre Specified Outcome: Change in Level of IGFBP2, IGFBP3 and Growth Hormone
Description: Serum samples and peripheral blood mononuclear cells (PBMNC) for pharmacodynamic activity with potential biomarkers for IMC-A12 (including, but not limited to: IGFBP2, IGFBP3 and Growth Hormone) obtained from optional blood specimens both before initiation of androgen deprivation therapy and twelve weeks after initiation of combined therapy. Results are reported as the difference between baseline and 12 weeks after start of therapy.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 18 | 9
pg/mL
  IGFBP-I | -946 (2309.3) | -904 (32362.4)
  IGFBP-III | 13893 (47335.2) | 291 (13344.5)
  GH | 66 (159.9) | -25 (327.8)

10. Other Pre Specified Outcome: Change in Level of Insulin
Description: Serum samples and peripheral blood mononuclear cells (PBMNC) for pharmacodynamic activity with potential biomarkers for IMC-A12 (insulin) obtained from optional blood specimens both before initiation of androgen deprivation therapy and twelve weeks after initiation of combined therapy. Results are reported as the difference between baseline and 12 weeks after start of therapy.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: ulU/mL
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Number analyzed (Participants) | 18 | 9
ulU/mL | 0 (5.1) | 0 (1.5)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: Participants were monitored for toxicity prior to each cycle or at more frequent intervals appropriate for that participant, as judged by the treating physician.
Arm/Group | Arm I (Androgen Deprivation and Cixutumumab) | Arm II (Androgen Deprivation Therapy)
Serious Adverse Events (participants affected / at risk) | 10/101 | 4/104
Other Adverse Events (participants affected / at risk) | 101/101 | 94/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Androgen Deprivation and Cixutumumab) (N=101) | Arm II (Androgen Deprivation Therapy) (N=104)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Death NOS (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Androgen Deprivation and Cixutumumab) (N=101) | Arm II (Androgen Deprivation Therapy) (N=104)
Anemia (Blood and lymphatic system disorders) | 39 | 30
Tinnitus (Ear and labyrinth disorders) | 6 | 1
Blurred vision (Eye disorders) | 11 | 4
Flashing lights (Eye disorders) | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 9
Constipation (Gastrointestinal disorders) | 17 | 9
Diarrhea (Gastrointestinal disorders) | 24 | 8
Dry mouth (Gastrointestinal disorders) | 10 | 1
Nausea (Gastrointestinal disorders) | 16 | 6
Oral pain (Gastrointestinal disorders) | 10 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5
Chills (General disorders) | 6 | 3
Edema limbs (General disorders) | 9 | 8
Fatigue (General disorders) | 66 | 47
Flu like symptoms (General disorders) | 9 | 0
Pain (General disorders) | 24 | 21
Urinary tract infection (Infections and infestations) | 6 | 2
Bruising (Injury, poisoning and procedural complications) | 10 | 1
Alanine aminotransferase increased (Investigations) | 19 | 14
Alkaline phosphatase increased (Investigations) | 10 | 16
Aspartate aminotransferase increased (Investigations) | 15 | 14
Blood bilirubin increased (Investigations) | 6 | 3
Creatinine increased (Investigations) | 24 | 12
Lymphocyte count decreased (Investigations) | 3 | 10
Neutrophil count decreased (Investigations) | 14 | 4
Platelet count decreased (Investigations) | 33 | 5
Weight gain (Investigations) | 4 | 7
Weight loss (Investigations) | 11 | 2
White blood cell decreased (Investigations) | 7 | 9
Anorexia (Metabolism and nutrition disorders) | 12 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 11 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 55 | 25
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 6
Hypokalemia (Metabolism and nutrition disorders) | 3 | 8
Hyponatremia (Metabolism and nutrition disorders) | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 9
Dizziness (Nervous system disorders) | 23 | 9
Dysgeusia (Nervous system disorders) | 13 | 0
Headache (Nervous system disorders) | 12 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 5
Anxiety (Psychiatric disorders) | 8 | 7
Depression (Psychiatric disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 8 | 10
Libido decreased (Psychiatric disorders) | 3 | 9
Hematuria (Renal and urinary disorders) | 10 | 6
Urinary frequency (Renal and urinary disorders) | 24 | 18
Urinary incontinence (Renal and urinary disorders) | 11 | 2
Urinary urgency (Renal and urinary disorders) | 6 | 4
Erectile dysfunction (Reproductive system and breast disorders) | 5 | 12
Pelvic pain (Reproductive system and breast disorders) | 8 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 21 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9 | 0
Hot flashes (Vascular disorders) | 49 | 69
Hypertension (Vascular disorders) | 27 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less